CLINICAL TRIAL: NCT07004933
Title: Rapid ART Initiation With BIC/FTC/TAF in HIV-infected People Who Inject Drugs (Naive or Re-linking to Care): a Pilot Study of an Integrated Care Model
Brief Title: Rapid Antiretroviral Treatment Initiation With BIC/FTC/TAF in HIV-infected People Who Inject Drugs (PWID)
Acronym: BFTAFDU
Status: Completed | Type: Observational
Sponsor: Hellenic Scientific Society for the Study of AIDS, Sexually Transmitted and Emerging Diseases (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: BFTAFDU-1
Record Dates: First submitted 2025-05-05; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: HIV Positive People Who Inject Drugs
MeSH Terms: interventions — bictegravir; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed- and re-linking to care previously- diagnosed HIV-positive subjects: HIV-positive PWID (people who inject drugs) subjects that enroll in the study within 7 days from the first visit in the clinic and are treatment-naïve or have discontinued antiretroviral treatment (ART) for more than 3 months from enrollment.
  Interventions: Drug: bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF)

INTERVENTIONS:
Drug: bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF) — Rapid antiretroviral treatment initiation with BIC/FTC/TAF

SUMMARY:
The goal of this clinical study is to evaluate the effectiveness, safety and patient experience of an integrated care pathway combining rapid antiretroviral (ART) initiation with BIC/FTC/TAF and peer navigation for treatment naïve newly-diagnosed or relinking HIV-infected PWIDs, in terms of viral suppression rates, adverse events and patient-reported health outcomes (PROs).

The main objectives of the study are the assessment of:

* The viral suppression rates at 24 weeks after the rapid initiation of ART with BIC/FTC/TAF coupled with secured peer-navigation in adult HIV-positive PWID who are treatment-naïve or re-linking to care
* The safety and tolerability of BIC/FTC/TAF in the specific context of rapid ART initiation in adult PWID who are treatment-naïve or re-linking to care from baseline until Week 24. Patients will receive their medication according to the standard of care and will visit the clinic as usual. No extra visits or extra lab tests will be performed.

DETAILED DESCRIPTION:
Taking into account the increased rates of new cases of HIV infection among people who inject drugs (PWID) in Greece, it is proposed the conduct of the observational study with the aim to assess whether clinical outcomes can be improved by the implementation of rapid ART initiation in newly diagnosed HIV-positive PWIDs and re-linking to care previously diagnosed HIV-positive PWIDs with a suitable medication, such as BIC/FTC/TAF, combined with peer-navigation support that can help the afflicted patients overcome social barriers and challenges. Therefore, this pilot study aims to evaluate the effectiveness, safety and patient experience of an integrated care pathway combining rapid ART initiation with BIC/FTC/TAF and peer navigation for treatment naïve newly-diagnosed or relinking HIV-infected PWIDs, in terms of viral suppression rates, adverse events and patient-reported health outcomes (PROs). Given the armamentarium of potent ART regimens, HIV infection has been transformed from a terminal illness into a chronic condition, thus, evaluating the impact of ARTs from patients' perspective is increasingly used [17]. The results of this study are expected to contribute towards informed health policy practices, accelerating and ameliorating care and providing the basis to curb the HIV epidemic and bringing us closer to its end.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female PWID subjects ≥18 years old
2. Documented and confirmed diagnosis of HIV infection
3. Naïve to ART or having discontinued ART for more than 3 months and relinking to care without documented resistance to any of the components of BIC/FTC/TAF or having missed more than once during the last 12 months, their monthly appointment for ART prescription renewal.
4. Willingness of patients to start OST or already being in OST.
5. Subjects willing and able to understand and provide written informed consent prior to participation in the study.
6. Females may be eligible for enrolment if they are i) of non-child-bearing potential or ii) if they are of child-bearing potential must have a negative pregnancy test at initial screening and agree to use throughout the study a medically acceptable method of contraception (barrier and/or hormonal method) or iii) are sterilized.

Exclusion Criteria:

1. Centers for Disease Control and Prevention Category C at baseline or presenting with clinical symptoms suggestive of opportunistic infections precluding rapid ART initiation per EACS guidelines 2020.
2. Alanine aminotransferase (ALT) >5 times upper limit normal (ULN) - Subjects with severe hepatic impairment (Child-Pugh score>9).
3. eGFR<30 ml/min
4. Any serious medical condition which would compromise the safety of the subject. Subject has a pre-existing mental, physical, or severe substance abuse disorder that may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations and assessments. Subject has a condition or disorder which may interfere with drug absorption or render the subject unable to take oral medication.
5. Subject is, in the opinion of the Investigator, unable to complete the study dosing period and protocol evaluations and assessments. Patients with alcohol and drug use problems that in the view of the Investigator will compromise participation in the study.
6. Subject has any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study. Any verified grade 4 abnormality would exclude a subject from participation in the study.
7. Subject is receiving or has received within 14 days prior to screening, any drug that has been classified as contraindicated from use with BIC/FTC/TAF
8. Pregnant or breast-feeding subjects.
9. Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-positive PWID subjects that enroll in the study within 7 days from the first visit in the clinic and are treatment-naïve or have discontinued antiretroviral treatment (ART) for more than 3 months from enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with a viral load of <50 copies/ml | Week 24 after treatment initiation
  The measurement is performed at Week 24 according to FDA snapshot analysis
The percentage of subjects experiencing a grade 3 or 4 adverse event | From baseline until Week 24 after treatment initiation
  The record of adverse events (related or not related to study treatment) grade 3 or 4

SECONDARY OUTCOMES:
The percentage of subjects with viral load <50 copies/ml at Week 48 | At Week 48 after treatment initiation
  The measurement is performed after Week 24 according to FDA snapshot analysis
The percentage of subjects with viral load <50 copies/ml other time points | At Weeks 4, 12, 24, 36, and 48 after treatment initiation
  The measurements are performed in several time points after treatment initiation
The difference in the percentage of subjects with a viral load of <50 copies/ml at Weeks 24 and 48 | At Week 24 and 48 after treatment initiation
  The difference in the percentage of subjects with a viral load of <50 copies/ml will be compared to a historic matched control group
The percentage of subjects experiencing a grade 3-4 adverse event after Week 24 | From Week 24 to Week 48 after treatment initiation
  The record of adverse events (related or not related to study treatment) grade 3 or 4 after Week 24
The mean change of CD4 count, CD4 (%) and CD4/CD8 ratio | From baseline to Week 48 after treatment initiation
  The evaluation of the change of CD4 count, CD4 (%) and CD4/CD8 ratio from treatment initiation to Week 48
The percentage of subjects retained in care at Weeks 24 and 48 | At Weeks 24 and 48, after treatment initiation
  The percentage of subjects that remain in the treatment at Weeks 24 and 48, after treatment initiation
The percentage of subjects lost to follow-up | From treatment initiation to Week 48
  The percentage of subjects that did not remain in the study until Week 48
The percentage of subjects with linkage and retention in OST programs | At Weeks 12, 24, and 48
  The monitoring of subjects that remained in the OST care until completion of Week 48, after treatment initiation.
The percentage of adherent patients during the study | At Weeks 4, 12, 24, 36, and 48
  Self-assessed adherence to study treatment at several time points during the study by using SMAQ questionnaire
The percentage of subjects with protocol-defined virologic failure at Week 12 and 24 | At Weeks 12 and 24, after treatment initiation
  The percentage of subjects with protocol-defined virologic failure i.e., plasma HIV-RNA >400 copies/ml at Week 12 confirmed on a second sample drawn 15-21 days later or 2 consecutive plasma HIV-RNA >50 copies/ml within 15-21days as of Week 24 at Week 12 and 24
The percentage of subjects requiring discontinuation/modification of treatment | From baseline to Week 48, after treatment initiation
  The percentage of subjects requiring discontinuation/modification of treatment with BIC/FTC/TAF throughout the study up to Week 48 due to: (i) Baseline resistance to one of the study drugs, and (ii) Adverse events.
The percentage of subjects harbouring a virus developing resistance | From the point of virological failure to Week 48
  The percentage of subjects harbouring a virus developing resistance associated mutations at the time of protocol-defined virological failure until Week 48
The percentage of subjects accepting initiation of ART and remaining in the study to Week 48 | From treatment initiation to Week 48
  The percentage of subjects 1) accepting initiation of ART within 7 days from first clinic visit through standard interview (according to EACS guidelines) and 2) accepting initiation of ART within 7 days from first clinic visit through standard interview (according to EACS guidelines) and remaining adherent to ART at Week 4, Week 12, Week 24, and Week 48.
The number and type of concomitant medications | From Day 0 to Week 48
  The number and type of concomitantly received medications from Day 0 and up to Week 48.
Changes in the scores of EuroQol Group 5-Dimension 3-Level (EQ-5D-3L) questionnaire | From baseline to Week 48
  The change in PRO scores EuroQol Group 5-Dimension 3-Level (EQ-5D-3L) from baseline at Weeks 4, 12, 24, 36, and 48. This evaluate the quality of life for several activities like mobility, self care etc. There is a scale from 0 to 100, 0 is for the worst health and 100 is for the best health.
Changes in the scores of HIV- Symptom Index (HIV-SI) questionnaire | From baseline to Week 48
  The HIV Symptom Index (HIV-SI) is a concise, validated questionnaire developed to assess overall symptom distress in people living with HIV, as well as to capture clinically relevant symptom clusters associated with the condition. Patient symptom distress is quantified by evaluating changes in Patient-Reported Outcome (PRO) scores derived from the HIV-SI, enabling effective monitoring of symptom burden over time.
Changes in the scores of Treatment Satisfaction Questionnaire for Medication (TSQM) | From baseline to Week 48
  The change in PRO scores in TSQM relative to Week 4 at Weeks 12, 24, 36, and 48. This questionnaire evaluates the level of satisfaction or dissatisfaction with the medication that a patient is taking during the clinical study. The scale is from 1 to 7, from extremely dissatisfied to extremely satisfied, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mina Psichogiou, Professor, Principal Investigator — General Hospital of Athens "LAIKO"
Locations (3):
- Greece (3):
  - General Hospital of Athens "EVAGGELISMOS", Athens, Attica
  - General Hospital of Athens "LAIKO", Athens, Attica
  - University General Hospital "ATTIKON", Athens, Attica

IPD SHARING:
Plan to Share IPD: Undecided
The decision is depending on the scope that the data will be asked - in case of an interested project, the request will be evaluated